CLINICAL TRIAL: NCT06691490
Title: Functional MRI Protocols for Studying the Neural Correlates of Effort Perception and the Effects of Targeted rTMS Protocols on Perceived Effort and Effort-based Decision-making
Brief Title: The Relationships Between Neural Correlates of Effort Perception and Physical Activity Engagement
Acronym: EffortLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: IRMage (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 38RC23.0416
Record Dates: First submitted 2024-11-07; First posted 2024-11-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: fMRI Research; Transcranial Magnetic Stimilation; EEG Brain Oscillations; Motor Task; Ischemic Nerve Block (INB); Muscle Vibration Protocol
Keywords: Perception of effort

STUDY DESIGN:
Intervention Model Description: Effort Perception; fMRI; EEG; Networks; Propioception
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation Sham (Experimental): Participants will engage in 4 cycling exercise visits and 4 effort-discounting task visits. Each of these 8 visits will be associated with one of the 4 stimulation conditions: vibration condition, sham vibration condition, cTBS over SMA. These 8 visits will be randomized across participant
  Interventions: Device: Transcranial Magnetic Stimulation Sham
- TMS (Placebo Comparator): cTBS over precuneus (control site).
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Sham — cTBS over SMA and cTBS over precuneus (control site)

SUMMARY:
Objectives and research hypothesis Physical inactivity is a major health concern that has been linked to a variety of chronic diseases, including obesity, diabetes, cancer, cardiovascular diseases, and mental disorders. Recent studies have shown that regular physical activity can decrease the risk of SARS-CoV-2 infection, and severe COVID-19 illnesses, as well as improve antibody response to vaccine. As such, the adoption of a physically active lifestyle carries potential health benefits and has even been referred to as a "miracle cure" by the Academy of Royal Medical Colleges. Despite the implementation of policies that aimed to encourage regular physical activity, the prevalence of insufficient physical activity in high-income countries has increased since 2001 (32% in 2001 vs. 37% in 2018). Given the limited impact of health policies on physical activity engagement, it is essential to explore other avenues of research that can contribute to understanding this high level of inactivity and driving innovative strategies for encouraging physical activity. In this context, the automatic attraction of individuals toward activities associated with low-effort exertion is thought to play a key role in physical inactivity. Physical activity involves exerting physical effort, i.e., intensifying physical energy to achieve certain goals, such as increasing the force to lift a heavy object. This physical intensification is associated with the phenomenological experience of energy exertion. Higher effort perception is thought to be aversively valued by inactive individuals, inhibiting their engagement in regular physical activity. However, there is a lack of knowledge regarding the neural correlates of effort perception and how they relate to physical inactivity. It is crucial to gain insights into these neural correlates, especially to enhance our comprehension of the significance of effort minimization in physical inactivity. This project aims to decrease effort perception and improve the valuation of effort, incentivize regular physical activity, and improve overall health outcomes.

Objective 1. Despite ongoing research, there is a lack of agreement on the neural mechanisms underlying effort perception as well as the role of sensorial feedback. Tasks EEG and fMRI aim to address this issue with original experimental methods in order to identify this neural mechanism.

Hypothesis 1. Following A) muscle vibration and B) Induced ischemic paralysis and anesthesia, we expect decreased effort perception associated with a lower cortical S1 activation, unchanged activation in premotor structures, and preserved functional connectivity between premotor regions and S1.

Objective 2. To unravel the neural interaction between efference copy and reafferent muscle spindle signals that contribute to effort perception Hypothesis 2. The neural correlates of effort perception involve interactions between premotor and sensory brain structures. Neural activation patterns of the brain regions implicated in effort perception vary depending on an individual's inclination to engage in physical activity.

Objective 3. Task 3 will examine the potential of non-invasive brain stimulation techniques (TMS) to reduce effort perception in turn increase its perceived value quantified with the CR100 scale, the outcome variable of this study.

Hypothesis 3. Vibration-induced desensitization of muscle spindles and the SMA cTBS reduce effort perception and improve the subjective value of physical effort.

DETAILED DESCRIPTION:
Our society is currently facing a pandemic of physical inactivity that is responsible for numerous chronic diseases and deaths. Despite the implementation of policies aimed at encouraging regular physical activity, the prevalence of physical inactivity remains high. It then seems necessary to explore other areas of research that could explain this level of inactivity and guide the implementation of new strategies to make the population more active. In this context, the tendency of most individuals to gravitate towards activities associated with a low perception of effort seems to play a central role in many barriers to engaging in physical activity. The perception of effort, which refers to the perception of the physical resources invested in a physical task, seems to be evaluated aversively by inactive individuals, limiting their engagement in physical activity. However, the neuropsychological bases of effort perception and how they are involved in physical inactivity remain poorly understood today. Therefore, clarifying the neural substrates involved in this perception and understanding how they determine engagement in physical activity is essential to help increase the population's level of physical activity. The hypothesis guiding this project is that reducing the perception of effort so that a particular intensity physical activity is perceived as less demanding facilitates engagement and the maintenance of a physically active lifestyle. In this context, the primary objective of this project will be to clarify the neural substrates involved in the perception of effort through a functional MRI study and to identify whether neuropsychological mechanisms related to the perception of effort differentiate individuals who have an aversion or an attraction to physical activity. Based on these results, the second objective will be to evaluate whether repetitive transcranial magnetic stimulation techniques targeting key nerve structures and reducing the perception of effort improve the value of effort and engagement in regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects all ranges age
* Exclusion Criteria:
* Neurologic conditions that may bias the EEG or fMRI results such as epilepsy, tumors; stroke; which can be a casual MRI finding during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Effort perception | From enrollment up to 12 months after
  Physical effort scale Category (C)-Ratio (R) (CR) scaling 100 or Borg centiMax® Scale (CR100) is a measure from 0 to 100 to rate the intensity of effort perception, where 0 means "nothing at all" (i.e. "no perception of effort at all") and 100 means "Maximal", that is, the maximal perception of effort experienced.

SECONDARY OUTCOMES:
Resting-state and task fMRI functional connectivity | From enrollment to 15 weeks after 60 healthy subjects will be assessed (4 subjects per week)
  Task fMRI condition A) induce ischemic paralysis and anesthesia: an MRI-compatible two chamber cuff will be placed over participants' upper arm outside the scanner and inflated to 250 mmHg until total abolishment of light touch sensation below the elbow is achieved46. This generally takes 20-40 min B) Task fMRI control condition. They will perform voluntary isometric handgrip contractions at moderate and strong perceived effort intensities based on the CR100 with their dominant hand. These two intensities were chosen to assess the impact of perceived effort level on brain activity, while avoiding excessive head movement that could occur at higher intensities and controlling for the development of neuromuscular fatigue C) Resting-state fMRI: 10-min resting-state fMRI scan to assess functional connectivity between different brain regions.
EEG event related synchronization | From enrollment to 40 weeks after
  ERSP analyses will allow us to examine changes in alpha (8-13 Hz) and beta (13-30 Hz) neural oscillations within predetermined regions of interest during spindle desensitization. This will be done trougth the application of vibration at the myotendinous junction of the biceps brachii using a custom-made vibrator. Following the successful methodology of the PI in PoC1 and 2, we will apply the vibration for a 10-min period with a frequency of 100 Hz and an amplitude of approximately 2 mm in the vibration condition.

CONTACTS AND LOCATIONS:
Overall Officials: Florian MONJO, Principal Investigator — Université de Chambéry
Locations (1):
- Plateforme IRMaGe, La Tronche, France

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in a secure server (NetExplorer, managed by the SFRI of the USMB). Access to the database will be limited with specific rights assigned to the different people involved in the project. Data extraction will automatically de-identified data
Supporting Information: Analytic Code
Time Frame: During the study
Access Criteria: Researchers and technicians involved in the project will have access to the data by a sharing lin
URL: https://www.netexplorer.fr/en/la-societe-netexplorer/

REFERENCES:
- [Background] Pageaux B. Perception of effort in Exercise Science: Definition, measurement and perspectives. Eur J Sport Sci. 2016 Nov;16(8):885-94. doi: 10.1080/17461391.2016.1188992. Epub 2016 May 30. PMID 27240002
- [Background] Inzlicht M, Shenhav A, Olivola CY. The Effort Paradox: Effort Is Both Costly and Valued. Trends Cogn Sci. 2018 Apr;22(4):337-349. doi: 10.1016/j.tics.2018.01.007. Epub 2018 Feb 21. PMID 29477776
- [Background] Hallam J, Jones T, Alley J, Kohut ML. Exercise after influenza or COVID-19 vaccination increases serum antibody without an increase in side effects. Brain Behav Immun. 2022 May;102:1-10. doi: 10.1016/j.bbi.2022.02.005. Epub 2022 Feb 5. PMID 35131444
- [Background] Christensen MS, Lundbye-Jensen J, Geertsen SS, Petersen TH, Paulson OB, Nielsen JB. Premotor cortex modulates somatosensory cortex during voluntary movements without proprioceptive feedback. Nat Neurosci. 2007 Apr;10(4):417-9. doi: 10.1038/nn1873. Epub 2007 Mar 18. PMID 17369825
- [Background] Cheval B, Sieber S, Maltagliati S, Millet GP, Formanek T, Chalabaev A, Cullati S, Boisgontier MP. Muscle strength is associated with COVID-19 hospitalization in adults 50 years of age or older. J Cachexia Sarcopenia Muscle. 2021 Oct;12(5):1136-1143. doi: 10.1002/jcsm.12738. Epub 2021 Aug 6. PMID 34363345
- [Background] Cheval B, Boisgontier MP. The Theory of Effort Minimization in Physical Activity. Exerc Sport Sci Rev. 2021 Jul 1;49(3):168-178. doi: 10.1249/JES.0000000000000252. PMID 34112744